CLINICAL TRIAL: NCT05824117
Title: Enhancing Educational and Vocational Recovery in Adolescents and Young Adults With Early Psychosis Through Supported Employment and Education (SEE): A Randomized Controlled Trial. Acronym: SEEearly
Brief Title: Enhancing Educational and Vocational Recovery in Adolescents and Young Adults With Early Psychosis Through Supported Employment and Education.
Acronym: SEEearly
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Prof. Dr. med. Andreas Bechdolf, Professor, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 470569697; DRKS00029660 (Registry Identifier: German Clinical Trials Register)
Record Dates: First submitted 2023-03-15; First posted 2023-04-21 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Persistent Delusional Disorder; Acute and Transient Psychotic Disorder, Unspecified; Schizophrenia; Schizoaffective Disorder; Other Nonorganic Psychotic Disorders; Unspecified Nonorganic Psychosis
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Mental Disorders | interventions — Palliative Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (TAU+SEE) (Experimental): The experimental intervention is treatment as usual (TAU) for adolescents and young adults with early psychosis in the respective recruitment centers for 12 months plus Supported Employment and Education following the Individual Placement and Support model.
  Interventions: Other: Individual Placement and Support (IPS)
- Control Group (TAU) (No Intervention): The control condition is treatment as usual (TAU) for adolescents and young adults with early psychosis in the respective recruitment centers for 12 months (including medical review, pharmacological treatment, and psychosocial support: group programs and social counseling to external government-funded vocational programs).

INTERVENTIONS:
Other: Individual Placement and Support (IPS) — IPS is an evidence-based practice for helping people with severe mental illness to gain and maintain competitive employment or/and mainstream education with nine well defined key principles that can be reliably assessed by the IPS Fidelity Scale for Young Adults.
  Interventions range from engagement techniques (i.e. motivational interviewing) to individualized education/employment searches and from experience-based educational/employment assessment to benefits in counseling/work incentives planning.
  Arms: Intervention Group (TAU+SEE)

SUMMARY:
Psychotic disorders often develop a chronic course with devastating consequences for individuals, families, and societies usually with first onset during adolescence and early adulthood. Early intervention programs, which provide intensive, phase specific, psychosocial, and pharmacological treatment for people in the first five years after the initial psychotic episode (early psychosis) can significantly improve the outcome and are therefore strongly recommended in national and international guidelines. However, most early intervention programs in people with early psychosis still focus on improving symptoms and relapse prevention, rather than targeting educational and vocational recovery, although engagement in work and education is a high priority for young people with early psychosis and reduces the social disability associated with the disorder. The aim of the present study is to explore the effects of Supported Employment and Education (SEE) following the Individual Placement and Support (IPS) model in people with early psychosis. The investigators compare treatment as usual (TAU) in an outpatient psychiatric setting to TAU plus SEE.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of early psychosis (DSM 5: schizophrenia spectrum and other psychotic disorders (297.1, 298.8, 295.4, 295.9, 295.7, 298.8, 298.9) within the last 5 years currently treated as outpatients
* sufficient linguistic and intellectual abilities to take part in the study
* interest in competitive employment or/and mainstream education
* written informed consent

Exclusion Criteria:

* Learning disability or mental retardation as well as insufficient German language abilities (< A2)
* physical or organic handicap that seriously impede work or educational functioning

Ages: 16 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 184 (Estimated)
Dates: Start 2022-10-18 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Primary outcome | 12 months
  The primary outcome is the binary indicator "Participating steadily for at least 50% of the 12 month follow-up in competitive employment or/and mainstream education". Days in competitive employment or/and mainstream education will be assessed monthly. Competitive employment is defined as jobs that anyone can apply for regardless of disability status. It comprises part and full-time positions, as well as seasonal or temporary positions depending upon the business needs of the employer. Mainstream education is defined in accordance with OECD as educational programs that are certificating or rather degree bearing and open to the general public.

SECONDARY OUTCOMES:
Length of competitive employment or/and mainstream education | 12 months
  Length of competitive employment or/and mainstream education (measured in days)
Time to first competitive job/mainstream education | 12 months
  Time to first competitive job/mainstream education (measured in days)
Monthly wages | 12 months
  Monthly wages (measured in Euro)
Educational attainment | 12 months
  Educational attainment (measured in degrees/qualifications and ECTS points per semester)
Social return on investment (SROI) | 12 months
  SROI will be computed as the ratio of 'benefits´ to 'total investment´ for each participant and is expressed as percentage. Participants' earnings in both competitive and non-competitive jobs, education, and apprenticeship hereby account as 'benefits´. 'Investments´ are defined as the total vocational program costs and total costs of mental health service per participant.
Subjective quality of life | 12 months
  Subjective quality of life will be measured with the World Health Organization Quality of Life-BREF, a short version of the World Health Organization Quality of Life 100 scale. It's a self-report questionnaire which assesses 4 domains of quality of life: physical health, psychological health, social relationships, and environment. Participants express how much they have experienced the items in the preceding 4 weeks on a 5-point Likert scale ranging from 1 (not at all) to 5 (completely).Higher scores indicate a better quality of life.
Psychopathology | 12 months
  Measured with the Positive and Negative Syndrome Scale (PANSS). The PANSS is a clinical interview rating the patient from 1 to 7 on 30 different symptoms. Ranges for the Positive Scale are 7 (minimum of symptoms) to 49 (maximum of symptoms), for the Negative Scale 7 (minimum of symptoms) to 49 (maximum of symptoms) and for the General Psychopathology Scale 16 (minimum of symptoms) to 112 (maximum of symptoms). Ratings are based on the interview as well as reports of family member and/or primary care workers. The interviewer must be trained to a standardized level of reliability.
General substance abuse | 12 months
  General substance abuse (mininum use of 3 times per week per substance) is measured by a modified version of the Addiction Severity Index (ASI).
Cannabis use | 12 months
  Cannabis use is specifically measured using the Daily Sessions, Frequency, Age of Onset and Quantity of Cannabis Use Inventory (DFAQ-CU).
Relapse | 12 months
  Assessed according to DSM 5 relapse definition criteria.
Hospitalization | 12 months
  Number of inpatient stays and duration of stays (measured in days) will be assessed.
Functional impairment | 12 months
  Functional impairment with regard to occupational activity and participation will be assessed using a short version of the International Classification of Functioning, Disability, and Health (Mini-ICF-APP) instrument. The instruments consists of 13 capacity dimensions: adherence to regulations, planning and structuring of tasks, flexibility, applying expertise, capacity to judge and decide, endurance, assertiveness, contacts with others, teamwork capacity, self-care, mobility, proactivity and familiar and intimate relationships. Each dimension is rated from 0 (no impairment) to 4 (full impairment).
Overall functional impairment | 12 months
  Overall level of functioning will be assessed using the Global Assessment of Functioning (GAF) scale. The GAF is a numeric scale to rate social, occupational and psychological functioning of an individual. Scores range from 1 (severely impaired) to 100 (extremely high functioning).

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Bechdolf, Prof., Principal Investigator — Klinik für Psychiatrie und Psychotherapie, Charite Universitätsmedizin Berlin
Locations (6):
- Germany (6):
  - Klinik für Sozialpsychiatrie, Zentrum für Psychiatrie Reichenau, Reichenau, Baden-Wurttemberg
  - Klinik für Psychiatrie und Psychotherapie, LMU Klinikum, München, Bavaria
  - Klinik für Psychiatrie, Psychotherapie und Psychosomatik II, Günzburg, Ulm, Bavaria
  - Klinik für Psychiatrie und Psychotherapie Charité Campus Mitte, Berlin
  - Klinik für Psychiatrie, Psychotherapie und Psychosomatik Vivantes Klinikum am Urban, Berlin
  - Klinik für Psychiatrie, Universitätsklinikum Hamburg Eppendorf, Hamburg

IPD SHARING:
Plan to Share IPD: No